CLINICAL TRIAL: NCT03933280
Title: Nalbuphine/Dexmedetomidine Versus Nalbuphine/Propofol Conscious Sedation for Cataract Extraction Under Topical Anaesthesia: A Double-Blind Randomized Trial
Brief Title: Conscious Sedation for Cataract Operations Under Topical Anaesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abd-Elazeem Abd-Elhameed Elbakry, Associate professor of anaesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019/3/25/9
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Nalbuphine; Propofol; Dexmedetomidine; benoxinate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: An independent anaesthesiologist not involved in the study will open the randomisation envelope just before the premedication and will prepare the appropriate drug-filled syringes according to the code and will not take part in the management and observations. (Syringes and infusion lines will be concealed by wrapping with an aluminium foil). A blinded investigator that will not be involved in the anaesthetic management of the patients, will collect the intra-operative and postoperative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): nalbuphine/propofol group
  Interventions: Drug: Nalbuphine; Drug: Propofol; Drug: Benoxinate Hydrochloride 0.4% Eye Drops
- Droup D (Active Comparator): Nalbuphine/dexmedetomidine group
  Interventions: Drug: Nalbuphine; Drug: Dexmedetomidine; Drug: Benoxinate Hydrochloride 0.4% Eye Drops

INTERVENTIONS:
Drug: Nalbuphine — i.v. nalbuphine bolus of 50 μg/kg.
  Other Names: Nalbuphine bolus
Drug: Propofol — A bolus i.v. dose of propofol 0.5 mg/kg followed by an infusion of 0.025 mg/kg/min
  Other Names: propofol infusion
  Arms: Group P
Drug: Dexmedetomidine — i.v. loading dose of dexmedetomidine 1 μg/kg over 10 min followed by a maintenance infusion of 0.5 μg/kg/h.
  Other Names: Dexmedetomidine infusion
  Arms: Droup D
Drug: Benoxinate Hydrochloride 0.4% Eye Drops — Benoxinate hydrochloride 0.4% eye drops instilled twice, 5 minutes apart.
  Other Names: Topical anaesthesia of the eye

SUMMARY:
Topical anaesthesia of the eye for ophthalmologic procedures avoids pain and discomfort of local anaesthetic injection in the peribulbar or retrobulbar block so that patient comfortability is achieved. Sedation during topical anaesthesia of the eye is mostly required to achieve anxiolysis, amnesia and keeping the patient calm all through the procedure. In the present study, the investigators will investigate the effect of nalbuphine/dexmedetomidine versus nalbuphine/propofol on the sedation as a primary outcome, intra-operative, postoperative analgesia, vital signs, patient and surgeon satisfaction and side effects as secondary outcomes

DETAILED DESCRIPTION:
In both groups, the patients will receive i.v. nalbuphine 50 μg/kg. Patients in group D, will receive an i.v. loading dose of dexmedetomidine 1 μg/kg over 10 min followed by a maintenance infusion of 0.5 μg/kg/h. Patients in group P, will receive a bolus i.v. dose of propofol 0.5 mg/kg followed by an infusion started at 0.025 mg/kg/min .If sedation score was <3, rescue sedation with boluses of midazolam 0.01 mg/kg will be given. If the patient complained of pain (Numerical verbal pain rating scale ≥3) during the surgery, i.v. fentanyl 50 μg will be given as an intra-operative rescue analgesic and the surgeon will be instructed to use additional topical local anaesthetic eye drops if appropriate. After the completion of surgery, all infusions will be stopped, and the patients will be shifted to the postanaesthetic care unit (PACU) to be monitored for 2 hours before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Both genders,
* 20 and 65 years,
* American Society of Anesthesiologists (ASA) physical status I and II,
* Scheduled for cataract extraction surgery under topical anaesthesia.

Exclusion Criteria:

* Known allergy to local anaesthetics,
* Allergy to study drugs,
* Second or third-degree heart block,
* Alcohol or drug abuse
* Morbid obesity, pregnant and lactating females,
* Patients with severe cardiac, renal and hepatic disorders.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Sedation score | perioperative
  The degree of sedation assessed by Ramsay sedation score(1 = anxious, agitated, restless;2 = cooperative, oriented, tranquil; 3 = responds to commands only; 4 = brisk response to light glabellar tap or loud noise; 5 = sluggish response to light glabellar tap or loud noise; 6 = no response), score of (1) means inadequate sedation. Score (2 to 4) indicates acceptable sedation. Score (5) or (6) excessive sedation.

SECONDARY OUTCOMES:
Heart rate | perioperative
  Heart rate in beats/minutes
Mean arterial blood pressure | perioperative
  Mean arterial blood pressure in mmHg
Oxygen saturation | perioperative
  Arterial oxygen saturation as a percentage of the total haemoglobin
Analgesia | perioperative
  Measured by Numerical Pain Rating scale where the patient verbally rates pain from 0 "no pain" to 10 "worst imaginable pain"

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, MD, Principal Investigator — Associate professor
Locations (1):
- Faculty of Medicine, Cairo, Shebin El-kom, Egypt